CLINICAL TRIAL: NCT05886686
Title: Validation of a Contactless Sensor for Measuring Vital Signs for Hospital Inpatients
Brief Title: Contactless Vital Signs Measurement Study (CVMS)
Acronym: CVMS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Melbourne Health (Other)
Responsible Party: Sponsor
Other Study IDs: RMH89542
Record Dates: First submitted 2023-03-21; First posted 2023-06-02 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-03

CONDITIONS: Vital Signs; Inpatients; Hospital-at-home
MeSH Terms: interventions — Thermometers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hospitalised inpatients: Ten patients admitted into the Acute Care of the Elderly (ACE) ward will be approached for inclusion in the study. Patients will be given written information about the trial. Nursing staff looking after these patients will be asked to utilise the device after vital sign measurements obtained from standard hospital equipment when conducting routine vital sign measurements. Nurses will do this for the duration of the admission of 7days, thus generating 28 paired data points for comparison.
  Interventions: Device: Validation of the accuracy of a combined oximeter, thermometer and heart rate measurement device
- Inpatients at home: Fifteen patients admitted into the home-based ward would be approached for inclusion in the study. Participants will undergo a 20 minute education session then be supplied with the device, companion app (user interface) on a mobile tablet, and written information about the trial.
  Participants will be asked to measure their vital signs four times a day, with one of those measurements occurring immediately after the clinical nurse' home review using standard hospital equipment for vital sign measurements (this matched pair of vital signs measurements will be taken as reference). Participants will do this for at least 7 days, thus generating 7 matched data points for comparison against reference, and 21 data points where participants independently conducted vital signs measurements with the Norbert sensor.
  Interventions: Device: Validation of the accuracy of a combined oximeter, thermometer and heart rate measurement device

INTERVENTIONS:
Device: Validation of the accuracy of a combined oximeter, thermometer and heart rate measurement device — Validation of the combined device measurements compared with standard of care devices

SUMMARY:
This study asks the question - Can vital signs be accurately measured via a contactless device and can this be independently done by inpatients in their homes? Primary objectives are to validate the accuracy of contactless vital sign measurements in comparison with vital signs measurements of heart rate, oxygen saturation, temperature using standard ward equipment (the reference standard).

DETAILED DESCRIPTION:
'Vital signs' such as heart rate (HR), temperature and peripheral blood oxygen saturation (SpO2) are routinely measured four times a day amongst hospitalised patients. However, this frequency of monitoring is unable to be replicated amongst patients in the RMH@Home Acute program. Also known as Hospital In The Home (HITH), RMH@Home Acute nurses and doctors deliver treatments to patients at home in substitution for a hospital admission. Home-based reviews are conducted one to two times daily, with more frequent reviews limited by travelling times and geographical constraints.

Accordingly, this study aims to investigate the accuracy and user-friendliness of new contactless technology to measure patients 'vital signs', paving the way towards enabling home-based patients to independently measure their vital signs during their admission. Besides enabling increased frequency of routine monitoring, this technology can also be applied to improve ad hoc assessments when patients report clinical concerns by enabling vital signs to be remotely measured by patients and/or their carers whilst clinicians travel to their homes to deliver treatment. Results from publication of this study will add to lexicon of knowledge regarding the utility of remote monitoring devices in monitoring and detecting clinical deterioration amongst hospitalized patients at home.

In this two-stage study, participants' vital signs obtained by the new contactless sensor are first compared with standard vital sign measurements obtained by nursing staff on the hospital ward. Should the sensor be found to obtain similar measurements thus indicating accuracy and feasibility of use amongst hospital patients, the second stage of this study involves investigating the feasibility of participants utilising these devices to measure their vital signs in the home-setting.

ELIGIBILITY:
Inclusion Criteria:

* Admitted inpatients within two hospital wards
* Patients expected to remain admitted within the two wards over 7 days of the study for availability of their vital sign measurements
* technological capability to utilise the device's companion app, as evidenced by ownership and utilisation of a 'smart' device (eg smartphone)

Exclusion Criteria:

* Cognitive disability impeding participants' ability to independently conduct vital sign measurements
* Clinical instability impeding participants' ability to independently conduct vital sign measurements
* Physical concerns (e.g. manual dexterity) impeding participants' ability to independently conduct vital sign measurements
* Environmental and technical issues such as lack of home Wi-Fi system, location of home in a 'Wi-Fi black spot', or unsafe home environments, that impede participants' ability to independently conduct vital sign measurements

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted patients that will require routine vital signs measurements with routine hospital equipment as part of standard of care; who will also be able to utilise a contactless vital sign measurement device at a matched timeframe to their routine vital signs measurements.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy validation - heart rate | 7 days
  Concordance of heart rate (beats per minute) measurements via the test device in comparison with nurse-conducted measurements of heart rate using standard ward equipment (reference standard). These measurements are deemed to be similar and acceptable for clinical purposes if within +/- 10% of the reference standard.
Accuracy validation - pulse oximetry for peripheral venous blood oxygen saturation | 7 days
  Concordance of pulse oximetry (percentage saturation) measurements via the test device in comparison with nurse-conducted pulse oximetry measurements of peripheral blood oxygen saturation using standard ward equipment (reference standard). These measurements are deemed to be similar and acceptable for clinical purposes if within +/- 10% of the reference standard.
Accuracy validation - temperature | 7 days
  Concordance of peripheral temperature (degree celsius) measurements via the test device in comparison with nurse-conducted temperature measurements using standard ward equipment (reference standard). These measurements are deemed to be similar and acceptable for clinical purposes if within +/- 10% of the reference standard.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Melbourne Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No